CLINICAL TRIAL: NCT04930692
Title: A Prospective Single-center Cohort Study "Preoperative Identification of Sentinel Lymph Nodes Using Contrast-enhanced CT Lymphography in Breast Cancer Patients"
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Saint Petersburg State University, Russia (Other)
Responsible Party: Principal Investigator, Ruslan Ahmedov, MD, Saint Petersburg State University, Russia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 03/21
Record Dates: First submitted 2021-06-10; First posted 2021-06-18 (Actual); Last update posted 2022-09-06 (Actual); Status verified 2022-09

CONDITIONS: Breast Neoplasms; Sentinel Lymph Node
Keywords: Breast cancer; Sentinel lymph nodes; CT-Lymphography
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Preoperative SLNs mapping provided by CT-lymphography method (Experimental): Sentinel lymph nodes will be mapped by contrast-enhanced CT lymphography in breast cancer patients. A mixture of 4 mL iopamidol and 2 mL of 1% lidocaine hydrochloride will be used as a contrast agent provided by periaoreolar injection. No later than 10 days after the CT lymphography patients will receive surgical treatment with sentinel lymph node biopsy using the ICG-fluorescence method.
  Interventions: Diagnostic Test: Contrast-enhanced CT lymphography with the periareolar injection of iopamidol

INTERVENTIONS:
Diagnostic Test: Contrast-enhanced CT lymphography with the periareolar injection of iopamidol — Patients who meet the inclusion/exclusion criteria will undergo the CT lymphography with periaoreolar injection of a mixture of 4 mL iopamidol and 2 mL of 1% lidocaine hydrochloride. Computed tomographic images will be obtained 1, 3, 5, and 10 minutes after administration of the iopamidol. Following enhancement of the lymphatic duct, the first lymph node to show enhancement will be defined as the SLN.
  No later than 10 days after the CT lymphography patients will receive surgical treatment. During breast cancer surgery identification of the SLN using the ICG-fluorescence method with injection of 2 ml indocyanine green into the skin of the areola and the biopsy of identified SLN will be performed. The comparison of the results of CT lymphography and SLN biopsy will be administrated by the investigator.

SUMMARY:
The main hypothesis of this study is that contrast-enhanced CT lymphography can be used for preoperative visualization of sentinel lymph nodes in breast cancer patients. We assume that CT lymphography is a high-sensitivity and high-specificity method for sentinel lymph nodes' mapping in breast cancer patients. We also assume that positive predictive value and negative predictive value for identification of presence or absence of metastases in sentinel lymph nodes (SLN) will be high enough for preoperative diagnosis of SLN metastases in breast cancer patients. This study will use CT lymphography with periareolar injection of iopamidol and standard protocols of sentinel lymph nodes biopsy using intraoperative indocyanine green (ICG) fluorescence.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years;
* Signed informed consent;
* Histologically confirmed breast cancer

Exclusion Criteria:

* Iodine allergy;
* Presence of distant metastases of breast cancer;
* Body mass index more than 40;
* Chronic cardiovascular and cerebrovascular diseases in the stage of decompensation or recent acute conditions (myocardial infarction, brain stroke, etc.)
* Suspected pregnancy;
* Severe hypothyroidism;
* Bronchial asthma in the stage of decompensation;
* Decompensated diabetes;
* Kidney or hepatic failure.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Estimated)
Dates: Start 2022-10-01 (Estimated); Primary Completion 2023-03-01 (Estimated); Study Completion 2023-08-01 (Estimated)

PRIMARY OUTCOMES:
Sensitivity and specificity of contrast-enhanced CT lymphography | 8 months
  First primary endpoint is to determine the sensitivity and specificity of contrast-enhanced CT lymphography for the preoperative detection of sentinel lymph nodes in breast cancer in comparison with the intraoperative fluorescence method.
Preoperative detection of sentinel lymph nodes metastases | 8 months
  Second primary endpoint is to assess the capabilities of contrast-enhanced CT lymphography for detecting metastases in sentinel lymph nodes in breast cancer patients

SECONDARY OUTCOMES:
Objective criteria for metastatic lesions of sentinel lymph nodes | 8 months
  Secondary endpoint is to identify objective criteria for metastatic lesions of sentinel lymph nodes (SLN), such as 1) the shape of the lymphatic duct; 2) the contrast enhancement of the SLN (full or heterogeneous); 3) the size of the SLN; 4) the form of the SLN; 5) the density of the SLN.

CONTACTS AND LOCATIONS:
Overall Officials: Ruslan Ahmedov, MD, Principal Investigator — Saint Petersburg State University Hospital
Locations (1):
- Saint-Petersburg State University Hospital, Saint Petersburg, Russia

IPD SHARING:
Plan to Share IPD: No